CLINICAL TRIAL: NCT02453113
Title: Immune-Related Trafficking and Signaling in Human Skin Associated With Low-Power, Infrared Laser Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Massachusetts General Hospital (Other); Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Kristen Kelly, M.D., Professor Departments of Dermatology and Surgery, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20151840
Record Dates: First submitted 2015-04-22; First posted 2015-05-25 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Vaccine Response Impaired
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- low power laser (Other): Signaling in Human Skin Associated with Low-Power, Infrared Laser Treatment
  Interventions: Other: low power laser

INTERVENTIONS:
Other: low power laser — Signaling in Human Skin Associated with Low-Power, Infrared Laser Treatment

SUMMARY:
The purpose of this is that the researcher can use low power Near Infrared laser treatment non-painful and non-damaging dose to changes the skin properties.The researcher can prove that signaling and a significant increase in the number of skin cells in skin tissue exposed to the laser can improve the human skin immune system to help improve human body response to vaccines.

DETAILED DESCRIPTION:
The researcher can use low power laser light one-minute exposures delivered to the skin at non-painful and non-damaging dose. The resulted in significant immunologic changes in the skin that included up-regulation of specific skin tissue and skin genes and the activation and mobilization of specific skin cells.

In the first part of the study, the researcher will make a determination of the laser irradiance that will be tolerated. The highest irradiance the subject tolerates for 1 minute will be identified as that subject's maximum tolerable irradiance. After all subjects are tested, researcher will select the highest irradiance that was tolerated and use this in the second phase of the study.

Approximately 24 hours after the first test exposures, each subject will receive a one minute laser treatment at the maximum tolerable irradiance. Four hours later, two skin biopsies will be collected from laser treated site a untreated.

One tissue sample will be test at UC Irvine Dept. of Dermatopathology to evaluate microscopic skin changes, one skin sample will be delivered to Massachusetts General Hospital to evaluate RNA and protein expression.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women with skin type 1 and 2
* Not pregnant

Exclusion Criteria:

* Use of systemic steroids, topical steroids, tanning solutions and anticoagulant
* History of HIV, mentally incompetent, prisoner, alcohol or drug impairment
* Abnormal photosensitivity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Kelly, MD, Principal Investigator — Beckman Laser Institute
Locations (2):
- United States (2):
  - Beckman Laser Institute, Irvine, California
  - Vaccine and Immunotherapy Center Massachusetts General Hospital, Charlestown, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Power Laser
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Low Power Laser
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 41 [18 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Skin Tissue Response to a Vaccine
Description: Change in inflammatory cells with low level laser will be measured.
Time Frame: up to 12 months
Population: We expect to demonstrate that the NIR laser dose elicits statistically significant dendritic cell trafficking to the human skin and induces cytokine/chemokine release and expression changes similar to that previously seen in mice.
Measure: Mean (Standard Error); unit: Total number of CD1a+ cells (5hpf)
Arm/Group | Low Power Laser
Number analyzed (Participants) | 10
Total number of CD1a+ cells (5hpf)
  Epidermis CD1a+ Langerhans cells Normal Control | 39.0 (1.6)
  Epidermis CD1a+ Langerhans cells Cases | 36.1 (1.6)
  Dermis CD1a+ Langerhans cells Normal Control | 21.5 (2.0)
  Dermis CD1a+ Langerhans cells Cases | 11.8 (1.6)
Statistical Analysis 1: Comparison: Low Power Laser; Test type: Superiority; The statistical end point of the study will be the changes in density of CD11c+ dermal dendritic cells between two biopsies from a study subject where one sample is subjected to laser irradiation and the other is the control. For assessment of statistical significance, we will apply a paired sample t-test

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Low Power Laser
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT02453113/Prot_SAP_ICF_000.pdf